CLINICAL TRIAL: NCT06879496
Title: Comparison of Oral Dexmedetomidine, Ketamine Versus Midazolam for Premedication in Children Undergoing Injuinal Surgeries
Acronym: CODKMPCIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed Zakarea Wfa, Associated professor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 36264PR1102/2/25
Record Dates: First submitted 2025-03-10; First posted 2025-03-17 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Pediatric; Anesthesia
Keywords: Ketamin; Midazolam; Dexmedetomidine; Oral; Pediatric
MeSH Terms: interventions — Midazolam; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group K (Active Comparator): Patients will receive orally ketamin 6 mg/kg.
  Interventions: Drug: Oral ketamin
- Group D (Active Comparator): Patients will receive orally dexmedetomidine 4 mcg kg -1
  Interventions: Drug: Oral dexmedetomidine
- Group M (Active Comparator): Patients will receive orally midazolam 0.5 mg kg -1.
  Interventions: Drug: Oral Midazolam

INTERVENTIONS:
Drug: Oral ketamin — Patients will be received oral ketamine before operation
  Arms: Group K
Drug: Oral Midazolam — Patients will be received oral Midazolam
  Arms: Group M
Drug: Oral dexmedetomidine — Patients will be received oral dexmedetomidine
  Arms: Group D

SUMMARY:
The aim of this study is to compare between oral dexmedetomidine, Ketamine or midazolam for premedication in children undergoing inguinal hernia surgeries.

DETAILED DESCRIPTION:
This randomized, double-blind comparative study will be carried out on 60 children undergoing inguinal hernia surgeries admitted to Tanta University Hospitals over a period from Mars 2025-September 2025.

An informed written consent will be obtained from the parents of these children. Every patient will receive an explanation of the purpose of the study and will have a secret code number.

Research results will be only used for scientific purpose. Any unexpected risk/s appearing during the course of research will be clarified to the participants and to the ethical committee on time.

Randomization and blinding:

Patients who meet the previous criteria will be enrolled in the study. Patients will be randomly classified into three equal groups: 20 patients will be enrolled in each group using computer generated random number in closed sealed, opaque envelopes:

(Group K): Patients will receive orally ketamin 6 mg/kg. (Group D): Patients will receive orally dexmedetomidine 4 mcg kg -1 (Group M): Patients will receive orally midazolam 0.5 mg kg -1. Patients and outcome assessors involved will be blinded to the study allocation and outcomes.

Study protocol:

Before operation, all patients will receive Groups M and D, K will receive an oral administration of 0.2 mg/kg of midazolam (up to a maximum of 15 mg) and 4 µg/kg of dexmedetomidine, 6mg ketamine respectively mixed with apple juice to make a final volume of 3-5 ml, in the preoperative holding area 40 min prior to anesthesia induction.

General anesthesia will be induced. Standard monitoring included electrocardiography (ECG), end-tidal carbon dioxide, arterial oxygen saturation continuously, pulse oximetry, and non-invasive BP every 5 min.

The anesthetic technique will be standardized in all patients. Anesthesia will be induced with sevoflurane 8% in oxygen 100% via a Jackson Rees breathing circuit. An i.v. cannula will be placed after induction of anesthesia. Patients then will receive i.v. propofol 1 mg kg-1 and a laryngeal Mask Airway will be applied.

Anesthesia will be maintained with sevoflurane in a 50% oxygen/air mixture. Spontaneous breathing will be maintained during the procedure. No other sedatives or opioids will be administered during the procedure. At the end of the procedure, the laryngeal mask will be removed, and the child will be transferred to the PACU once the airway will be maintained spontaneously and there will be no hemodynamic instability.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 3-7 years.
* Both sexes.
* American society of anesthesiologists (ASA) physical status (I-II).

Exclusion Criteria:

* Parents refusal.
* Patients with known allergy to the study drugs.
* Significant organ dysfunction.
* Cardiac dysrhythmia.
* Use of psychotropic medication, and mental retardation.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-09-10 (Actual); Study Completion 2025-09-10 (Actual)

PRIMARY OUTCOMES:
Primary outcome | on arrival in the operating room 30 min after end of study drug administration.
  five-point sedation score

SECONDARY OUTCOMES:
Secondary outcome | Till 1 hour after operation
  FLACC score Postoperative face, legs, activity, cry, and consolability (FLACC) scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed Zakarea Wfa, Tanta, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided